CLINICAL TRIAL: NCT07242716
Title: Evaluation of the Effect of Different Thread Designs on Primary Stability of Dental Implant Using Osseodensification Technique in Posterior Maxilla : Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Akram Osman, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: stability of dental implant
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Primary Stability of Knife Threads Dental Implant Versus Double Threads Using Osseodensification Technique
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knife threads design dental implant (Experimental): the intervention group is the knife threads dental implant using the osseodensification technique
  Interventions: Device: dental implant
- double threads design dental implant (Active Comparator): the control group is the double threads dental implant using osseodensification technique
  Interventions: Device: dental implant

INTERVENTIONS:
Device: dental implant — dental implant with double thread design
  Arms: double threads design dental implant
Device: dental implant — dental implant with knife threads design
  Arms: knife threads design dental implant

SUMMARY:
the aim of this study is to compare the primary stability of dental implant with knife threads design versus dental implant with double threads design using osseodensification technique in posterior maxilla .

DETAILED DESCRIPTION:
Introduction:

1. Background and rationale:

   Research question:

   Is the use of knife threads dental implants enhancing primary stability in the posterior maxilla more than double threads when using the osseodensification technique?

   Statement of the problem:

   Implant design affects implant stability especially thread design. Osseodensification (OD) working in a non-subtractive fashion, condense the implant osteotomy soft bone in lateral direction, leading to a greater bone volume and density, an increase in the bone implant contact, with subsequent increase in insertion torque levels, and reduction in micromotion (Seo et al., 2022). However, it has been claimed that OD increases the implant bone bed density but does not improve implant primary stability (Almutairi et al., 2018).

   Thus, the aim of this study is to evaluate the effect of different threads design on primary stability of dental implant using osseodensification on posterior edentulous maxillary region.
2. Rationale for conducting the research:

Dental implants have become a treatment option widely used for the replacement of lost teeth. The development of dental implants has had a major impact on the patients. The implant supported oral restoration has become an increasingly used treatment option for partially and completely edentulous patients (Duong et al., 2022).

The replacement of a tooth using an implant is derived from an evolution in concepts, technology, and clinical applications, following years of basic research and fundamental studies on the concept of osseointegration (Cooper and Shirazi, 2021).

Implant design parameters lay the foundation for properties like implant primary stability and ability to sustain loading during or after osseointegration (Huang et al., 2023). Implant design is divided into two major categories: micro design and macro design. Macro design includes implant body shape, thread and thread design, while micro design constitutes surface morphology, implant materials, and surface coating (Kumar et al., 2024).

Surgical techniques of implant placement also play a vital role in establishing osseointegration. If, during ostetomy preparation, drilling temperature exceeds 47°C for more than a minute, local osteonecrosis and impair osseointegration may happen (Soldatos et al., 2022).Various drilling protocols have been established for implant placement namely, conventional, under preparation or OD techniques (Inchingolo et al., 2021).

Therefore, a high initial (primary) implant stability is essential for successful osseointegration of implants with the adjacent bone, and this itself is influenced by several factors including implant design, size, macro-and micro-surface, quality and quantity of bone, and the surgical technique used for implant placement in addition to the operator's skills (Xiao et al., 2024).

Bone density is a key factor to consider when predicting implant stability. A good surgical technique and good stability favors implant osseointegration. The long-term success of implant therapy is achieved by the primary stability of the implant for mechanical support from the surrounding bone in the early stage and osseointegration between the surrounding bone and implant through bone regeneration and remodeling in the late stage (Huang et al., 2023). Primary stability is especially necessary in poor quality bone. The instability of dental implants results in fibrous encapsulation and failure to achieve osseointegration (Hossain et al., 2023).

Clinically, the dental implant primary stability can be evaluated using several techniques, such as the amount of torque needed during insertion, or after insertion using the resonance frequency analysis technology implemented in the Osstell device, or the mechanical percussion principle used in the Periotest (Almutairi et al., 2018).

Although the OD may minimize the use of other more invasive techniques, such as ridge splitting, sinus lifting, and onlay bone grafting, there has been a claim that the OD surgical technique may not be effective in improving the primary stability of dental implants, and that the dental implant macro-design is not crucial for the implant primary stability so long as the surrounding bone is of good quantity and quality (Othman et al., 2024).

Explanation for choice of comparators:

The use of osseodensification in combination with these thread designs is an important factor in this study, as it enhances bone density and improves implant stability through controlled bone compaction. Therefore, comparing different thread designs such as those with aggressive threads for great mechanical retention versus those with more moderate threads for less bone stress allows us to observe differences in primary stability outcomes.

7. Objectives: The aim of this study is to compare the primary stability of dental implant with knife threads design versus dental implant with double threads design using osseodensification technique.

Hypothesis:

We hypothesis that using knife threads dental implant will provide primary stability of dental implants in the posterior maxillary region more than double threads dental implant.

ELIGIBILITY:
Inclusion Criteria:

* age from 20 to 60 years
* both sex
* patient with deficient width in posterior maxilla

Exclusion Criteria:

* inadequate oral hygiene
* smoking habit > 10 cigarettes per day
* abuse of alcohol or drugs
* pregnancy
* local or systemic infection
* sever hepatic or renal dysfunction
* bony or soft tissue pathological condition at surgical site
* uncontrolled systemic diseases
* parafunctional habits
* inability or unwillingness to return for follow-up visits

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
primary stability of dental implant | primary stability will be measured immediately after implant placement and 2nd record after 4 months
  measuring the primary stability using osstell device and smart peg

SECONDARY OUTCOMES:
marginal bone height changes | after 6 months of dental implant placement
  measuring changes in marginal bone height using cone beam CT

IPD SHARING:
Plan to Share IPD: Undecided